CLINICAL TRIAL: NCT03984539
Title: A Randomized Controlled Trial of the Effectiveness of CBT-T vs CBT-E in a Community Clinic of Individuals With Eating Disorders
Brief Title: Comparing CBT-T to CBT-E in Non-low-weight Adults With Eating Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6278
Record Dates: First submitted 2019-05-29; First posted 2019-06-13 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-03

CONDITIONS: Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial comparing the efficacy of two outpatient psychological treatments for eating disorders that primarily differ in length. Investigators will use a longitudinal design that includes both interview and questionnaire measures to assess eating disorder symptoms and other mental health-related outcomes.
Who Masked: Outcomes Assessor
Masking Description: At the beginning of client's appointments with the staff psychometrist, patients will be reminded of the study, provided information about the study and asked if to participate in the study. If interest is indicated, then the psychometrist will thoroughly review the letter of information with patients. If patients agree to participate and sign the consent form, study measures will be given. The psychometrist will then inform their assigned therapist that the client wishes to participate in the study. To ensure the psychometrist is not aware of randomization, Philip Masson (study PI) will randomize the client to one of the two interventions using the website random.org. Philip Masson will inform the therapist of the randomization, and the therapist will then proceed with the appropriate treatment intervention. The PI will then keep track of randomization assignment in a separate excel file that the psychometrist does not have access to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-E (Active Comparator): Participants will be randomly assigned to one of two conditions (CBT-E or CBT-T). CBT-E will occur over the course of 25 weeks and be delivered as it typically is in the clinic setting of the investigators.
  Interventions: Behavioral: Cognitive Behavioural Therapy-Enhanced
- CBT-T (Experimental): Participants will be randomly assigned to one of two conditions (CBT-E or CBT-T). Participants who agree to participate will receive 10 weeks of CBT-T.
  Interventions: Behavioral: Cognitive Behavioural Therapy-Ten

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy-Enhanced — CBT-E is a 20-session transdiagnostic eating disorders treatment based on the principles of cognitive behavioural therapy which has been developed over the past 40 years. The treatment focusses on tracking and modifying eating behaviours, providing psychoeducation, addressing overvaluation of weight and shape, body image, food restriction and restraint, emotion regulation, and relapse prevention.
  Arms: CBT-E
Behavioral: Cognitive Behavioural Therapy-Ten — CBT-T is a 10-session treatment based on cognitive behavioural therapy. It was developed based on clinical experience as well as core components of evidence-based versions of CBT for eating disorders, including CBT-E. The aim of the intervention is to provide only the hypothesized critical elements of CBT for eating disorders so that the interventions can be provided quicker.
  Arms: CBT-T

SUMMARY:
Eating disorders are a difficult to treat illness with significant psychological and physical sequelae. Cognitive behavioural therapy (CBT) has been the most researched and supported intervention for eating disorders. A particular version of CBT for eating disorders, CBT-E (Fairburn, 2008), has been the focus of much research over the past decade. Despite promising results from initial CBT-E trials these findings have not always replicated well and evidence points to high drop-out in real-world settings. Further, CBT-E is a resource-intensive intervention, which may contribute to poorer access to care. In an attempt to overcome some of these barriers related to CBT-E, Waller and colleagues (2018) recently developed a brief (10 session) version of CBT for non-low-weight eating disorders (e.g., bulimia nervosa and binge eating disorder), referred to as CBT-T. Preliminary evidence from a case series of adult patients suggests that CBT-T has similar efficacy to CBT-E with low rates of drop-out. However, further evaluation of this brief treatment is needed, including direct comparisons with CBT-E. Indeed, given that no comparison group was included in the initial case series, it is unknown whether either CBT-T or CBT-E may be superior to the other. Thus, the aim of the current project is to examine CBT-T's efficacy in comparison to CBT-E as it has been implemented at the eating disorders service at London Health Science's Centre, and to determine whether either intervention is superior based on treatment outcome and treatment drop-out. Non-low-weight individuals with eating disorders assessed at the Adult Eating Disorders Service will be eligible to participate in the study. The principle investigator is Dr. Philip Masson, Ph.D., C. Psych., 519-685-8500 ext. 74866.

DETAILED DESCRIPTION:
Design:

As CBT-T is anticipated to achieve faster improvement, due to its brief nature, than CBT-E this research study is not utilizing a non-inferiority design. That is, differences between the two interventions are anticipated, at least initially. Over time, the two interventions may become similar in some aspects (final remission rate for completers) but not others (final remission rate utilizing intention to treat).

Hypotheses:

CBT-T will produce higher rates of symptom abstinence initially as the treatment takes approximately half as long as CBT-E and then at post-treatment follow-ups that effect will disappear using completer analysis. However, as drop-out is expected to be lower in CBT-T it is expected that CBT-T will consistently produce superior results to CBT-E with intention to treat analysis.

Recruitment:

Individuals who have been assessed at the Adult Eating Disorders Service and meet eligibility criteria will be informed by the assessor that they are eligible to participate in a trial examining a new treatment. The assessor will provide the letter of information for the study and the study will be explained to the participants and any questions the participants have about the study will be addressed. The assessor will inform the staff psychometrist at the service that the participant is eligible to participate in the study. Participants will be asked to participate in the study once the participants name has reached the top of the treatment waitlist and a clinician is able to see them. Once the patient's name reaches the top of the treatment wait-list the participant will meet with the psychometrist in preparation for treatment, as part of routine procedure, and asked to participate in the study. Due to the significant waiting list (currently 5-6 months) as well as the tendency for some clients to end up not accessing care, study participation will be sought when it is most relevant.

At the beginning of client's appointments with the staff psychometrist, patients will be reminded of the study, provided information about the study and asked if to participate in the study. If they indicate interest in participating, then the psychometrist will thoroughly review the letter of information with patients. If patients agree to participate and sign the consent form, study measures will be given. The psychometrist will then inform the assigned therapist that the client wishes to participate in the study. To ensure the psychometrist is not aware of randomization, Philip Masson (study PI) will randomize the client to one of the two interventions using the website random.org. Philip Masson will inform the therapist of the randomization, and the therapist will then proceed with the appropriate treatment intervention. The PI will then keep track of randomization assignment in a separate excel file that the psychometrist does not have access to. If clients do not wish to participate in the study, clients will be assessed using the clinic's standard program evaluation protocol and will receive treatment as usual (CBT-E). Once individuals are participating in the study only the assigned treatment will be received and this process will be clearly explained to participants. Participants can withdraw from the study at any time at which point their data collection would stop; however, participants would continue to receive their assigned treatment. If participants wish to end treatment, then participants will be able to reapply to the service after a 2-month waiting period, which is standard practice for the service.

Interventions:

CBT-E is a transdiagnostic eating disorders treatment based on the principles of cognitive behavioural therapy which has been developed over the past 40 years. The treatment focusses on tracking and modifying eating behaviours, providing psychoeducation, addressing overvaluation of weight and shape, body image, food restriction and restraint, emotion regulation, and relapse prevention. For non-low-weight individuals, the treatment is designed as a 21 session treatment (one orientation meeting and 20 treatment sessions). The adult eating disorders service has been utilizing this treatment approach on an outpatient basis for the past two years. All staff members have reviewed the reading material associated with the treatment, participated in online training for CBT-E and participate in weekly peer supervisions sessions where staff members support one another in utilization of the treatment. Therapists are encouraged to review relevant sections of the therapist manual as needed. The treatment is adhered to the manual as close as possible except for one major exception. In CBT-E the treatment is designed to be delivered twice weekly for the first 4 hours. Instead, the service provides weekly sessions as the patients and staff found it too difficult to make twice weekly sessions fit into their schedule. After approximately 17 weekly sessions then sessions drop down to every other week.

CBT-T is a 10-session treatment based on cognitive behavioural therapy. It was developed based on clinical experience as well as core components of evidence-based versions of CBT for eating disorders, including CBT-E. The aim of the intervention is to provide only the hypothesized critical elements of CBT for eating disorders so that the interventions can be provided quicker. As rapid response to treatment in CBT for eating disorders has been shown to be a key predictor of outcome, it is possible that a briefer intervention may not be necessarily less effective. Further, briefer interventions may result in reduced drop-out which would allow more clients to fully access treatment. The key elements of this intervention are similar to CBT-E except there is a less explicit focus on emotion regulation and the psychoeducation is provided in the moment as opposed to being provided as a separate element of treatment. Further, in CBT-T treatment is initially only offered for four sessions and then extended only if the patient is actively engaging in treatment, which is similar to the session 8 progress review in CBT-E but occurs earlier and is framed differently. The therapy is delivered using a session by session checklist of core tasks to facilitate adherence. The clinicians at the service will receive training in CBT-T in the form of an 8-hour workshop delivered by one of the creators of the intervention, Glenn Waller. Further, the treatment manual will also be provided to all clinicians and read prior to the workshop. The clinicians will also participate in group supervision for one hour per week focusing on effective delivery of CBT-T.

Data Analysis:

Data will be analyzed using SPSS (version 24). Treatment groups will be compared on baseline characteristics (e.g., eating disorder symptoms) using independent samples t-tests and chi-square for categorical measures. Percentage scores will be calculated to determine attrition rates at each stage of treatment and chi-square analyses will be used to compare attrition/drop-out between the two treatment conditions. A two-level hierarchical linear model will be used to examine the influence of the intervention on change in symptoms over time. Level 1 (within-subjects) will include repeated measures of the dependent variable (e.g., EDE-Q scores, ED symptoms) and level 2 (between-subjects) will include treatment condition (CBT-T or CBT-E) and the interaction between condition and time. Separate models will be conducted for different outcome variables of interest. Both an intention to treat and completer analyses will be performed. For the intention to treat analysis multiple imputation will be utilized to handle the resultant missing data.

Power analyses: In accordance with recommendations for pilot RCTs by Rounsaville, Carroll, & Onken (2001), the investigators aim to have at least 20 participants per group (after attrition). Based on power analyses for repeated measures analysis of variance (ANOVA) for between-within group differences using G*power 3, a total sample size of 40 would yield >80% power to detect medium effects (f2 >.20), which represents a conservative approach, given increased power of multilevel modeling over traditional repeated measures ANOVA. Based on prior studies of CBT-T, the investigators anticipate an overall attrition rate of approximately 30%; thus, they propose to enroll 60 participants (30 per treatment condition) to detect an attrition-adjusted medium effect.

ELIGIBILITY:
Inclusion Criteria:

1. Non-underweight (BMI > 19) adults (aged > 17 years)
2. Diagnosis of bulimia nervosa (BN), binge eating disorder (BED), or otherwise specified feeding or eating disorder (e.g., subthreshold BN, subthreshold BED, purging disorder)

Exclusion Criteria:

1. Imminent risk for suicide
2. Profound cognitive impairment
3. Limited English language ability

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in the frequency of Binge Eating | Will be assessed Pre-Treatment; Post-Treatment (On average 10 weeks for CBT-T and 25 weeks for CBT-E), 3, 6, 12, 24 months post treatment. Treatment is on Average 10 weeks for CBT-T and 25 weeks for CBT-E
  Assessed using EDE (Fairburn, Cooper, & O'Connor, 2008) objective binge eating frequency for past month. Clients can answer anywhere from 0 binges to an infinite number of binges.
Change in the frequency of Vomiting | Pre-Treatment; Post-Treatment (On average 10 weeks for CBT-T and 25 weeks for CBT-E) 3, 6, 12, 24 months post treatment. Treatment is on Average 10 weeks for CBT-T and 25 weeks for CBT-E
  Assessed using EDE (Fairburn, Cooper, & O'Connor, 2008) vomiting frequency for past month. Clients can answer anywhere from 0 vomiting episodes to an infinite number of vomiting episodes.
Change in Eating Disorder Cognitions | Pre-Treatment; Post-Treatment (On average 10 weeks for CBT-T and 25 weeks for CBT-E), 3, 6, 12, 24 months post treatment. Treatment is on Average 10 weeks for CBT-T and 25 weeks for CBT-E
  Assessed using EDE-Q (Fairburn & Beglin, 2008) Global Score. Lowest possible global score is 0 and highest possible global score is 6. The higher the score the more severe the eating disorder cognitions.

SECONDARY OUTCOMES:
Binge Eating Change over the Course of Treatment | Pre-treatment and weekly while receiving treatment. Once a week for up to 10 weeks of treatment for CBT-T and up to 25 weeks of treatment for CBT-E.
  Binge eating symptoms recorded weekly via the Eating Disorder-15 (Tatham et al., 2015). Clients will indicate frequency of binging on this measure. The higher the number the more often clients are binging. Binge eating frequency is not part of a scale rather, the number indicated represents the number of binges clients report having.
Vomiting Change over the Course of Treatment | Pre-treatment and weekly while receiving treatment. Once a week for up to 10 weeks of treatment for CBT-T and up to 25 weeks of treatment for CBT-E.
  Vomiting symptoms recorded weekly via the Eating Disorder-15 (Tatham et al., 2015). The higher the number the more often clients are vomiting. Vomiting frequency is not part of a scale rather, the number indicated represents the number of vomiting episodes clients report having.
Working Alliance change over the Course of Treatment | Pre-treatment and weekly while receiving treatment. Once a week for up to 10 weeks of treatment for CBT-T and up to 25 weeks of treatment for CBT-E.
  Working alliance as measured by the Working Alliance Short-Form (Hatcher & Gillaspy, 2006). Each item is rated on a 1-7 scale, where 1 = 'Not at all', and 7 = 'Completely'. The highest possible score is 84 and the lowest possible score is 12. The higher the score the better working alliance towards therapist and client.
Change in Depression symptoms | Pre-Treatment; Post-Treatment (On average 10 weeks for CBT-T and 25 weeks for CBT-E), 3, 6, 12, 24 months post treatment. Treatment is on Average 10 weeks for CBT-T and 25 weeks for CBT-E
  Assess via the Patient Health Questionnaire (PHQ-9; Kroenke, Spitzer, & Williams, 2001). The highest possible score is 27 and the lowest possible score is 0. The lower the score the less depression symptoms.
Change in anxiety symptoms | Pre-Treatment; Post-Treatment (On average 10 weeks for CBT-T and 25 weeks for CBT-E), 3, 6, 12, 24 months post treatment. Treatment is on Average 10 weeks for CBT-T and 25 weeks for CBT-E
  Assess via the Generalized Anxiety Disorder Questionnaire (Spitzer, Kroenke, Williams, & Lowe, 2006). The highest possible score is 21 and the lowest possible score is 0. The lower the score the less anxiety symptoms.
Change in Loss of Control over Eating | Pre-Treatment; Post-Treatment (On average 10 weeks for CBT-T and 25 weeks for CBT-E), 3, 6, 12, 24 months post treatment. Treatment is on Average 10 weeks for CBT-T and 25 weeks for CBT-E
  Assessed using the Loss of Control over Eating Scale-Brief (LOCES-B; Latner et al., 2014). The brief version of the LOCES is a 7-item measure used to assess severity of loss of control over eating. Example items include "I continued to eat past the point when I wanted to stop" and "I felt I could not do anything other than eat." Items are scored on 5-point Likert scale ranging from 1=never to 5=Always. 7 is the lowest possible score and 35 is the highest possible score. The lower the score the better as this indicates better control over eating. The higher the score the worse as this indicates the inability to control eating.
Change in Motivation | Pre-Treatment; Post-Treatment (On average 10 weeks for CBT-T and 25 weeks for CBT-E), 3, 6, 12, 24 months post treatment. Treatment is on Average 10 weeks for CBT-T and 25 weeks for CBT-E
  Assessed via the Readiness and Motivation Questionnaire (Geller et al., 2013). Overall scores can be calculated to determine precontemplation, action, internality, and confidence for changing symptoms. Scores range from 0% to 100%, where higher scores indicate more of the construct.
Change in Impulsivity | Pre-Treatment; Post-Treatment (On average 10 weeks for CBT-T and 25 weeks for CBT-E), 3, 6, 12, 24 months post treatment. Treatment is on Average 10 weeks for CBT-T and 25 weeks for CBT-E
  Assessed via the the negative urgency scale (from the full version of the UPPS-P). Ranges from 1 strongly agree, 2 somewhat agree, 3 Disagree and 4 Disagree Strongly. 12 is the lowest possible score and 44 is the highest possible score. The lower the score the better as this indicates less impulsivity. The higher the score the worse, as this indicates high impulsivity.
Change in overall perceived quality of life | Pre-Treatment; Post-Treatment (On average 10 weeks for CBT-T and 25 weeks for CBT-E), 3, 6, 12, 24 months post treatment. Treatment is on Average 10 weeks for CBT-T and 25 weeks for CBT-E
  Assessed via the world health organization quality of life scale-brief (WHOQOL-BREF). The WHOQOL-BREF produces a quality of life profile. It is possible to derive 4 domains. 2 items are examined separately- question 1 asks about an individuals overall perception of quality of life and question 2 asks about an individuals overall perception of their health. The 4 domain scores denote an individuals perception of quality of life in each particular domain. Domain scores are scaled in a positive direction (higher scores denote higher quality of life). The mean score of items within each domain is used to calculate the domain score. Mean scores are then multiplied by 4 in order to make domain scores comparable with the scores in the WHOQOL-100 (full version of the scale).

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Phoenix, Principal Investigator — London Health Sciences Centre
Locations (1):
- The Adult Eating Disorders Service, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berg KC, Peterson CB, Frazier P, Crow SJ. Psychometric evaluation of the eating disorder examination and eating disorder examination-questionnaire: a systematic review of the literature. Int J Eat Disord. 2012 Apr;45(3):428-38. doi: 10.1002/eat.20931. Epub 2011 Jul 8. PMID 21744375
- [Background] Butler, A. C., Beck, A. T., & Cohen, L. H. (2007). The personality belief questionnaire-short form: Development and preliminary findings. Cognitive Therapy and Research, 31, 357-370. http://dx.doi.org/10.1007/s10608-006-9041-x
- [Background] Byrne SM, Fursland A, Allen KL, Watson H. The effectiveness of enhanced cognitive behavioural therapy for eating disorders: an open trial. Behav Res Ther. 2011 Apr;49(4):219-26. doi: 10.1016/j.brat.2011.01.006. Epub 2011 Jan 27. PMID 21345418
- [Background] Cyders MA, Littlefield AK, Coffey S, Karyadi KA. Examination of a short English version of the UPPS-P Impulsive Behavior Scale. Addict Behav. 2014 Sep;39(9):1372-6. doi: 10.1016/j.addbeh.2014.02.013. Epub 2014 Mar 3. PMID 24636739
- [Background] Dear BF, Titov N, Sunderland M, McMillan D, Anderson T, Lorian C, Robinson E. Psychometric comparison of the generalized anxiety disorder scale-7 and the Penn State Worry Questionnaire for measuring response during treatment of generalised anxiety disorder. Cogn Behav Ther. 2011;40(3):216-27. doi: 10.1080/16506073.2011.582138. Epub 2011 Jul 20. PMID 21770844
- [Background] Fairburn, C. G. (2008). Cognitive behavior therapy and eating disorders. New York, NY: Guilford.
- [Background] Fairburn, C. G., & Beglin, S. J. (2008) Eating Disorder Examination Questionnaire (6.0). In Fairburn CG. Cognitive Behavior Therapy and Eating Disorders. New York: Guilford Press.
- [Background] Fairburn, C. G., Cooper, Z., & O'Connor, M. (2008). Eating Disorder Examination (16.0D). In Fairburn C. G., Cognitive Behavior Therapy and Eating Disorders. New York: Guilford Press.
- [Background] Fairburn CG, Cooper Z, Doll HA, O'Connor ME, Bohn K, Hawker DM, Wales JA, Palmer RL. Transdiagnostic cognitive-behavioral therapy for patients with eating disorders: a two-site trial with 60-week follow-up. Am J Psychiatry. 2009 Mar;166(3):311-9. doi: 10.1176/appi.ajp.2008.08040608. Epub 2008 Dec 15. PMID 19074978
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G*Power 3.1: tests for correlation and regression analyses. Behav Res Methods. 2009 Nov;41(4):1149-60. doi: 10.3758/BRM.41.4.1149. PMID 19897823
- [Background] Geller J, Brown KE, Srikameswaran S, Piper W, Dunn EC. The psychometric properties of the Readiness and Motivation Questionnaire: a symptom-specific measure of readiness for change in the eating disorders. Psychol Assess. 2013 Sep;25(3):759-768. doi: 10.1037/a0032539. Epub 2013 May 6. PMID 23647034
- [Background] Hatcher, R. L., & Gillaspy, J. A. (2006). Development and validation of a revised short version of the working alliance inventory. Psychotherapy Research, 16, 12-25. http://dx.doi.org/10.1080/10503300500352500
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Latner JD, Mond JM, Kelly MC, Haynes SN, Hay PJ. The Loss of Control Over Eating Scale: development and psychometric evaluation. Int J Eat Disord. 2014 Sep;47(6):647-59. doi: 10.1002/eat.22296. Epub 2014 May 26. PMID 24862351
- [Background] Lowe B, Unutzer J, Callahan CM, Perkins AJ, Kroenke K. Monitoring depression treatment outcomes with the patient health questionnaire-9. Med Care. 2004 Dec;42(12):1194-201. doi: 10.1097/00005650-200412000-00006. PMID 15550799
- [Background] Moriarty AS, Gilbody S, McMillan D, Manea L. Screening and case finding for major depressive disorder using the Patient Health Questionnaire (PHQ-9): a meta-analysis. Gen Hosp Psychiatry. 2015 Nov-Dec;37(6):567-76. doi: 10.1016/j.genhosppsych.2015.06.012. Epub 2015 Jun 18. PMID 26195347
- [Background] Newman, M., Zuellig, A. R., Kachin, K. E., Constanitno, M. J., Przeworski, A., Erickson, T., & Cashman-McGrath, L. (2002). Preliminary reliability and validity of the generalized anxiety disorder questionnaire-IV: A revised self-report diagnostic measure of generalized anxiety disorder. Behavior Therapy, 33, 215-233. https://doi.org/10.1016/S0005-7894(02)80026-0
- [Background] 2024 exceptional surveillance of eating disorders: recognition and treatment (NICE guideline NG69) [Internet]. London: National Institute for Health and Care Excellence (NICE); 2024 May 15. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK607987/ PMID 39405396
- [Background] Paap D, Dijkstra PU. Working Alliance Inventory-Short Form Revised. J Physiother. 2017 Apr;63(2):118. doi: 10.1016/j.jphys.2017.01.001. Epub 2017 Feb 21. No abstract available. PMID 28336298
- [Background] Pellizzer ML, Waller G, Wade TD. Body image flexibility: A predictor and moderator of outcome in transdiagnostic outpatient eating disorder treatment. Int J Eat Disord. 2018 Apr;51(4):368-372. doi: 10.1002/eat.22842. Epub 2018 Feb 19. PMID 29457252
- [Background] Rounsaville BJ, Carroll KM, Onken LS. A stage model of behavioral therapies research: Getting started and moving on from stage I. Clinical Psychology: Science and Practice. 2001;8(2):133-142.
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Tatham M, Turner H, Mountford VA, Tritt A, Dyas R, Waller G. Development, psychometric properties and preliminary clinical validation of a brief, session-by-session measure of eating disorder cognitions and behaviors: The ED-15. Int J Eat Disord. 2015 Nov;48(7):1005-15. doi: 10.1002/eat.22430. Epub 2015 May 26. PMID 26011054
- [Background] Turner H, Marshall E, Wood F, Stopa L, Waller G. CBT for eating disorders: The impact of early changes in eating pathology on later changes in personality pathology, anxiety and depression. Behav Res Ther. 2016 Feb;77:1-6. doi: 10.1016/j.brat.2015.11.011. Epub 2015 Dec 1. PMID 26690743
- [Background] Waller G, Tatham M, Turner H, Mountford VA, Bennetts A, Bramwell K, Dodd J, Ingram L. A 10-session cognitive-behavioral therapy (CBT-T) for eating disorders: Outcomes from a case series of nonunderweight adult patients. Int J Eat Disord. 2018 Mar;51(3):262-269. doi: 10.1002/eat.22837. Epub 2018 Feb 8. PMID 29417603
- [Background] Wonderlich SA, Peterson CB, Crosby RD, Smith TL, Klein MH, Mitchell JE, Crow SJ. A randomized controlled comparison of integrative cognitive-affective therapy (ICAT) and enhanced cognitive-behavioral therapy (CBT-E) for bulimia nervosa. Psychol Med. 2014 Feb;44(3):543-53. doi: 10.1017/S0033291713001098. Epub 2013 May 23. PMID 23701891
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712